CLINICAL TRIAL: NCT05518487
Title: Safety and Immunogenicity of a Dose of the Sanofi-GSK Monovalent (B.1.351) CoV2 preS dTM-AS03 COVID-19 Vaccine in Kidney Transplant Recipients With a Persistently Low SARS CoV-2 Antibody Titer (COVID19-TB-04)
Brief Title: COVID Protection After Transplant - Sanofi GSK (CPAT-SG) Study
Acronym: CPAT-SG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: PPD Development, LP (Industry); Johns Hopkins University (Other); Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DAIT COVID19-TB-04
Record Dates: First submitted 2022-08-18; First posted 2022-08-26 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: COVID-19; Kidney Transplant
Keywords: Kidney transplant; COVID-19; Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Kidney transplant recipients (Experimental): This single-arm trial will administer a single dose of the Sanofi-GSK monovalent (B.1.351) CoV2 preS dTM-AS03 COVID-19 vaccine to kidney transplant recipients who demonstrate a persistently low (≤ 2500 u/mL) anti-spike antibody response after completion of primary series and bivalent booster of either the Moderna COVID-19 Vaccine or the Pfizer-BioNTech Vaccine, as described in their respective Food and Drug Administration (FDA) Emergency Use Authorizations (EUAs)
  Interventions: Biological: Sanofi-GSK monovalent (B.1.351) CoV2 preS dTM-AS03 COVID-19 vaccine

INTERVENTIONS:
Biological: Sanofi-GSK monovalent (B.1.351) CoV2 preS dTM-AS03 COVID-19 vaccine — 0.5 mL per dose of the Sanofi-GSK COVID-19 Vaccine will be administered intramuscularly in the deltoid muscle of the upper arm

SUMMARY:
An open label, non-randomized pilot study in kidney transplant recipients who received a completed primary series and bivalent booster of mRNA based COVID-19 vaccine and have ≤2500 U/mL SARS-CoV-2 S antibody concentration using the Roche Elecsys(R) anti-RBD assay. Up to 80 participants will be enrolled in this study. Eligible participants will receive a dose of the Sanofi-GSK monovalent (B.1.351) CoV2 preS dTM-AS03 COVID-19 vaccine candidate..

The primary objective is to determine whether a booster dose of the Sanofi-GSK monovalent (B.1.351) CoV2 preS dTM-AS03 COVID-19 vaccine will elicit an increased SARS-CoV-2 antibody response in participants who have failed to maintain an antibody titer >2500 U/mL (using the Roche Elecsys(R) anti-RBD assay) to 2 or more doses of mRNA based COVID-19 vaccine

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and provide informed consent
2. Individual ≥ 18 years of age.
3. Recipient of kidney transplant ≥12 months prior to enrollment, without treated allograft rejection in the 6 months preceding enrollment
4. Maintenance immunosuppressive regimen consisting of CNI and mycophenolate mofetil or mycophenolate, with or without ≤ 5mg/day prednisone or equivalent
5. Received completed primary series (3 doses) of mRNA vaccine (either the Moderna COVID-19 vaccine or Pfizer-BioNTech COVID-19 vaccine) as specified in the respective package inserts
6. Receipt a COVID-19 bivalent mRNA booster (Moderna or Pfizer-BioNTech) >30 days prior to enrollment.
7. Serum antibody titer up to 2500 U/mL at ≥ 30 days from the last dose of mRNA COVID-19 vaccine and

   * 30 days following receipt of a monoclonal antibody product or convalescent plasma for COVID-19, measured using the Roche Elecsys(R) anti-SARS-CoV-2 S assay
8. Platelet count greater than 30,000/cu mm must be confirmed in participants with a known history of bleeding disorder or thrombocytopenia (platelet count <50,000/cu mm)
9. A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

   1. Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year or surgically sterile

      OR
   2. Is of childbearing potential and agrees to use an effective contraceptive method or abstinence for 12 weeks post vaccine and while taking mycophenolate mofetil/mycophenolic acid

Exclusion Criteria:

1. Recipient of any number of doses of any COVID vaccine product other than the Moderna COVID-19 vaccine or the Pfizer-BioNTech COVID-19 vaccine
2. Recipient of any organ other than a kidney
3. Known current or prior Donor Specific Antibody (DSA)
4. Any change in transplant immunosuppression regimen (drug or dose) in response to suspected or proven rejection within the last 6 months
5. Known diagnosis of COVID-19 since last antibody test
6. Receipt of a monoclonal antibody product or convalescent plasma within the last 30 days
7. Known history of hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to a vaccine containing any of the same substances. (components listed in Section 6, and the CoV2 and AS03 Investigator's Brochure)
8. Bleeding disorder, or receipt of anticoagulants in the past 21 days preceding inclusion, contraindicating intramuscular (IM) vaccination based on Investigator's judgment
9. Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
10. Receipt of any vaccine in the 30 days preceding the study vaccine or planned vaccines in the 30 days following the study vaccine
11. Estimated Glomerular Filtration Rate <30mL/min/1.73m^2
12. Receipt of any cellular depleting agent (e.g. Antithymocyte globulin (ATG), Rituximab, Alemtuzumab, Cyclophosphamide) within 12 months preceding enrollment
13. Receiving systemic immunomodulatory medication(s) for any condition other than transplant
14. Any uncontrolled active infection
15. Infection with human immunodeficiency virus (HIV)
16. Maintenance immunosuppressive regimen that includes anything other than a CNI, mycophenolate/mycophenolate mofetil, and ≤ 5mg/day prednisone or equivalent
17. Recent (within one year) or ongoing treatment for malignancy, except for definitive surgical treatment of localized skin cancers
18. Any unstable acute or chronic illness, treatments, or findings which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the c candidate's ability to comply with study requirements or may impact the quality or interpretation of the data obtained from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorry Segev, MD, Ph.D., Study Chair — New York University Langone Health-Transplantation; Peter S Heeger, MD, Study Chair — Icahn School of Medicine at Mount Sinai: Transplantation; Christian P. Larsen, MD, D.Phil., Study Chair — Emory University School of Medicine: Transplantation; William A. Werbel, MD, Study Chair — Johns Hopkins University; Christine Durand, MD, Principal Investigator — Johns Hopkins University
Locations (6):
- United States (6):
  - University of California San Diego Medical Center: Transplantation, San Diego, California
  - UCSF School of Medicine: Transplantation, San Francisco, California
  - Emory University School of Medicine: Transplantation, Atlanta, Georgia
  - University of Illinois Medical Center: Transplantation, Chicago, Illinois
  - Johns Hopkins Institute for Clinical and Translational Research: Broadway Adult Outpatient Clinical Research Unit, Baltimore, Maryland
  - University of Wisconsin School of Medicine and Public Health: Transplantation, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait

RESULTS

PARTICIPANT FLOW:
Groups:
- SARS CoV-2 Anti-RBD Persistently Low: Kidney transplant recipients who have failed to maintain an antibody titer >2500 U/ml (using the Roche Elecsys® anti-RBD assay) to a completed primary series and bivalent booster of mRNA based COVID-19 vaccine
Period: Overall Study
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Started | 15
Completed | 12
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [54 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Years Since Transplant [Median (Inter-Quartile Range); unit: years] | 5.1 [3.1 to 8.1]
Number of Prior COVID-19 Vaccines Received [Count of Participants; unit: Participants]
  Four | 1
  Five | 11
  Six | 3
Days Between Last Vaccination and Antibody Screening [Median (Inter-Quartile Range); unit: days] | 222.5 [161 to 279]
Baseline SARS-CoV-2 Antibody Level [Median (Inter-Quartile Range); unit: U/mL] — Population: One participant vaccinated on study was subsequently discovered to have an inaccurate baseline antibody level of ≥ 2500 U/ml (2948.5 U/ml). This participant was excluded from the immunogenicity population for the primary endpoint as well as the corresponding baseline population.
  U/mL
    number analyzed (Participants) | 14
    (all) | 223.5 [53 to 934.5]

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants Who Reach a SARS-CoV-2 S Antibody Level >5000 U/mL
Description: The antibody is measured by using the Roche Elecsys(R) anti-RBD assay
Time Frame: At 30 days following a dose of vaccine
Population: 1 participant received study vaccine but was excluded from primary immunogenicity population; baseline SARS-CoV-2 was initially misreported as eligible (≤ 2500 U/ml). This patient is included in the demographics/baseline description population and in non-immunogenicity clinical or safety outcomes (e.g. death, graft loss, need for dialysis, acute rejection).
Measure: Count of Participants; unit: Participants
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 14
Participants | 0

2. Secondary Outcome: Composite That Includes Death, Graft Loss, Need for Dialysis, and Acute Rejection
Time Frame: Within 30 days following the study dose of vaccine
Population: Safety Population: Participant receiving study vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 15
Participants | 0

3. Secondary Outcome: Death
Time Frame: Within 30 days or within 60 days of the study dose of vaccine
Population: Safety population (Participant receiving study vaccine). 1 participant terminated the study after day 30. This patient who terminated prior to evaluation at 60 days had not had the 'event' at the time of termination and was censored.
Measure: Count of Participants; unit: Participants
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 15
Participants
  Death within 30 days of vaccine | 0
  Death within 60 days of vaccine: number analyzed (Participants) | 14
  Death within 60 days of vaccine | 0

4. Secondary Outcome: Graft Loss
Time Frame: Within 30 days or within 60 days of the study dose of vaccine
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 15
Participants
  Graft loss within 30 days of vaccine | 0
  Graft loss within 60 days of vaccine: number analyzed (Participants) | 14
  Graft loss within 60 days of vaccine | 0

5. Secondary Outcome: Need for Dialysis
Time Frame: Within 30 days or within 60 days of the study dose of vaccine
Population: Safety population (Participant receiving study vaccine) 1 participant terminated the study after day 30. This patient who terminated prior to evaluation at 60 days had not had the 'event' at the time of termination and was censored.
Measure: Count of Participants; unit: Participants
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 15
Participants
  Need for dialysis within 30 days of vaccine | 0
  Need for dialysis within 60 days of vaccine: number analyzed (Participants) | 14
  Need for dialysis within 60 days of vaccine | 0

6. Secondary Outcome: Acute Rejection
Time Frame: Within 30 days or within 60 days of the study dose of vaccine
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 15
Participants
  Within 30 days | 0
  Within 60 days: number analyzed (Participants) | 14
  Within 60 days | 0

7. Secondary Outcome: Local Vaccine Reactogenicity
Time Frame: Collected for 7 days following the study dose of vaccine)
Measure: Count of Participants; unit: Participants
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 15
Participants
  Injection Site Pain: Grade 0 (None) | 3
  Injection Site Pain: Grade 1 (Mild) | 11
  Injection Site Pain: Grade 2 (Moderate) | 1
  Redness: Grade 0 (None) | 14
  Redness: Grade 1 (Mild) | 0
  Redness: Grade 2 (Moderate) | 1
  Swelling: Grade 0 (None) | 14
  Swelling: Grade 1 (Mild) | 0
  Swelling: Grade 2 (Moderate) | 1

8. Secondary Outcome: Systemic Vaccine Reactogenicity
Time Frame: Collected for 7 days following the study dose of vaccine)
Measure: Count of Participants; unit: Participants
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 15
Participants
  Fever: Grade 0 (None) | 15
  Fever: Grade 1 (Mild) | 0
  Fever: Grade 2 (Moderate) | 0
  Headache: Grade 0 (None) | 14
  Headache: Grade 1 (Mild) | 0
  Headache: Grade 2 (Moderate) | 1
  Tired: Grade 0 (None) | 10
  Tired: Grade 1 (Mild) | 4
  Tired: Grade 2 (Moderate) | 1
  Muscle Pain: Grade 0 (None) | 14
  Muscle Pain: Grade 1 (Mild) | 0
  Muscle Pain: Grade 2 (Moderate) | 1
  Joint Pain: Grade 0 (None) | 13
  Joint Pain: Grade 1 (Mild) | 1
  Joint Pain: Grade 2 (Moderate) | 1
  Chills: Grade 0 (None) | 13
  Chills: Grade 1 (Mild) | 1
  Chills: Grade 2 (Moderate) | 1

9. Secondary Outcome: Adverse Events of Special Interest (AESIs), Including Potential Immune Mediated Diseases
Description: The categories of AESI that required special reporting in this protocol were: Anaphylactic reactions; Generalized convulsion; Thrombocytopenia; Thrombosis with thrombocytopenia syndrome; Myocarditis; Pericarditis; Potential immune-mediated diseases (pIMDs)
Time Frame: 1 year following the study dose of vaccine
Population: Safety Population (includes all subjects, including all follow-up for the 1 participant who decided to terminate early, and the 1 participant whose baseline antibody titer was misreported, and thus enrolled despite having an ineligible baseline antibody titer > 2500 U/ml).
Measure: Count of Participants; unit: Participants
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 15
Participants
  Experienced AESI | 0
  Did not experience AESI | 15

10. Secondary Outcome: Treated Acute Cell-mediated Allograft Rejection (Clinical or Biopsy-proven)
Time Frame: Within 60 days following the study dose of vaccine
Population: Safety Population. 1 participant terminated the study after day 30, prior to 60 day follow-up. One participant decided to terminate the study after day 30, prior to 90 days assessment; this participant had not experienced clinical or biopsy-proven rejection at any time prior to termination.
Measure: Count of Participants; unit: Participants
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 14
Participants | 0

11. Secondary Outcome: Treated Antibody-mediated Allograft Rejection (Clinical or Biopsy-proven)
Time Frame: Within 60 days following the study dose of vaccine
Population: Safety population (Participant receiving study vaccine). 1 participant terminated the study after day 30, prior to 60-day follow-up. One participant decided to terminate the study after day 30, prior to 60 days assessment; this participant had not experienced clinical or biopsy-proven anitbody-mediated rejection at any time prior to termination.
Measure: Count of Participants; unit: Participants
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 14
Participants | 0

12. Secondary Outcome: Development of de Novo Donor-specific Anti-human Leukocyte Antigens (HLA) Antibody
Time Frame: Within 90 days of the vaccine and up to 12-months post vaccine
Population: Safety population (Participant receiving study vaccine). 3 participants terminated the study prior to 1 year (1 after day 30, 2 after day 90). One participant decided to terminate the study after day 30, prior to 90 day or 1 year assessments; this participant had not experienced clinical or biopsy-proven anitbody-mediated rejection at any time prior to termination.
Measure: Count of Participants; unit: Participants
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 14
Participants
  Development within 90 days of vaccine | 0
  Development within 1 year of vaccine | 0

13. Secondary Outcome: Change in Pre-existing Donor-specific Anti-human Leukocyte Antigens (HLA) Antibody
Time Frame: From study entry to 90 days post vaccine and up to 12-months post vaccine
Population: Safety population (Participant receiving study vaccine). 3 participants terminated the study prior to 1 year (1 after day 30, 2 after day 90). One participant decided to terminate the study after day 30, prior to 90 day or 1 year assessments; this participant had not experienced clinical or biopsy-proven antibody-mediated rejection at any time prior to termination.
Measure: Count of Participants; unit: Participants
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 14
Participants
  to 90 days post vaccine | 0
  to 1 year post vaccine | 0

14. Secondary Outcome: Anti-RBD Antibody Concentration
Description: The antibody is measured by using the Roche Elecsys(R) anti-RBD assay
Time Frame: At 30 days after the study dose of vaccine
Population: Immunogenicity population (Participant receiving study vaccine, with baseline SARS-CoV-2 S anti-RBD assay ≤ 2500 U/ml). 1 participant received study vaccine but was excluded from immunogenicity population; baseline SARS-CoV-2 was initially misreported as eligible.
Measure: Median (Inter-Quartile Range); unit: U/ml
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 14
U/ml | 565 [153 to 2038]

15. Secondary Outcome: Fold Rise (FR) in Anti-RBD Antibody Concentration
Description: The Fold Rise is the dimensionless ratio between each participant's day 30 antibody titer (in U/ml) and the participant's baseline antibody titer (in U/ml) antibody is the antibody titers are measured by using the Roche Elecsys(R) anti-RBD assay.
Time Frame: From baseline to 30 days after the study dose of vaccine
Population: 1 participant received study vaccine but was excluded from immunogenicity population; baseline SARS-CoV-2 was initially misreported as eligible (≤ 2500 U/ml).
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 14
ratio | 1.8 [1.2 to 3.4]

16. Secondary Outcome: Monogram Pseudovirus Antibody Titers
Description: For selected variants of concern (prototype (Wuhan), beta, and omicron BA.1; additional alternative strains to be determined based on assay availability). tests unable to be performed
Time Frame: At 14 and 30 days after the study vaccine dose
Population: Data were not collected because tests were unable to be performed. Study funding was unexpectedly terminated prior to assessment of the samples. The assessment of these samples is not expected to be performed in the future.
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 0

17. Secondary Outcome: Median Range of Fold Rise (FR) in Monogram Pseudovirus Antibody Titers
Description: For selected variants of concern (prototype (Wuhan), beta, and omicron BA.1; additional alternative strains to be determined based on assay availability)
Time Frame: From baseline to 14 and 30 days after the study vaccine dose
Population: as for outcome 16
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year following the study dose of vaccine (See additional relevant information about adverse event collection in the Adverse Event Reporting Description).
Description: Time frame for All-Cause mortality: up to 1 year following the study dose of vaccine.
  Time frame for SAEs and AESIs: up to 1 year following the study dose of vaccine. For this study, AESIs are the following: Anaphylactic reactions; Generalized convulsion; Thrombocytopenia; Thrombosis with thrombocytopenia syndrome; Myocarditis; Pericarditis; or potential Immune-Mediated Diseases (pIMD).
  Time frame for non-serious AEs: up to 30 days following the study dose of vaccine.
Arm/Group | SARS CoV-2 Anti-RBD Persistently Low
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SARS CoV-2 Anti-RBD Persistently Low (N=15)
COVID-19 infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SARS CoV-2 Anti-RBD Persistently Low (N=15)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
WBC disorder (Blood and lymphatic system disorders) | 3 (3)
Hyperglycaemia (Endocrine disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Coronavirus infection (Infections and infestations) | 2 (2)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Haemoglobin increased (Investigations) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Contusion (Vascular disorders) | 1 (1)
Dizziness (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT05518487/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/87/NCT05518487/ICF_001.pdf